CLINICAL TRIAL: NCT02384837
Title: Effect of TCFA on Neointimal Coverage After EXCEL Biodegradable Polymer-coated Sirolimus-eluting Stents Implantation at 9 Months Follow-up: Evaluated by Optical Coherence Tomography and Fractional Flow Reserve
Brief Title: Effect of TCFA on Neointimal Coverage After PCI at 9 Months Follow-up
Status: Completed | Type: Observational
Sponsor: General Hospital of Chinese Armed Police Forces (Other)
Responsible Party: Sponsor
Other Study IDs: Effect of TCFA
Record Dates: First submitted 2014-12-25; First posted 2015-03-10 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2015-01

CONDITIONS: Unrecognized Condition
Keywords: national Cather Lad; Interventional Imaging Training Base

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- TCFA: EXCEL biodegradable polymer-coated sirolimus-eluting stent was implanted on lesions which include TCFA (>=1)
  Interventions: Device: EXCEL biodegradable polymer-coated sirolimus-eluting stent
- NO-TCFA: EXCEL biodegradable polymer-coated sirolimus-eluting stent was implanted on lesions which is not include TCFA
  Interventions: Device: EXCEL biodegradable polymer-coated sirolimus-eluting stent

INTERVENTIONS:
Device: EXCEL biodegradable polymer-coated sirolimus-eluting stent

SUMMARY:
Although drug-eluting stents have reduced rates of restenosis and late lumen loss compared with bare metal stents, late stent thrombosis (LST), a life-threatening complication of this technology, has emerged as a major concern. Researches indicated incomplete neointimal coverage of stent struts as the most important morphometric predictor of LST. Pathological research showed stenting disruption of adjacent vulnerable plaques can precipitate LST, Meanwhile, thin-cap fibroatheromas (TCFA) as the most important predictor of Major Adverse Cardiovascular. Therefore, there is a hypothesis that TCFA may impair intimal healing which are prone to LST in vivo.

Optical coherence tomography (OCT)is a high-resolution (<10 µm), catheter-based imaging modality capable of investigating detailed coronary plaque morphology in vivo.This study aimed to observe that TCFA will arise what of the effect on intimal healing of stent struts on the lesions which fractional flow reserve (FFR)≤0.75 after EXCEL biodegradable polymer-coated sirolimus-eluting stent was implanted at 9 months follow up: evaluated by OCT and FFR

DETAILED DESCRIPTION:
The primary end point is to Neointimal coverage after 9 months of the stent implantation.

Quality assurance plan that addresses data validation and registry procedures, including any plans for site monitoring and auditing.

Data checks to compare data entered into the registry against predefined rules for range or consistency with other data fields in the registry.

Source data verification to assess the accuracy, completeness, or representativeness of registry data by comparing the data to external data sources (e.g., medical records, paper or electronic case report forms, or interactive voice response systems).

Data dictionary that contains detailed descriptions of each variable used by the registry, including the source of the variable, coding information if used and normal ranges if relevant.

Standard Operating Procedures to address registry operations and analysis activities, such as patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management.

Sample size assessment to specify the number of participants or participant years necessary to demonstrate an effect.

ELIGIBILITY:
Inclusion Criteria:

* 18yrs≤Age≤75yrs
* stability and unstable angina pectoris (AP), chronic myocardial infarction (OMI) or confirmed myocardial ischemia
* De novo lesion at native coronary artery(Up to two target lesions)
* Lesion length ≤32mm
* RVD 2.5mm～4.0mm
* DS%≥70% by visual test
* Coronary artery bypass surgery (coronary artery bypass grafting) patients
* Subjects are willing to follow the specified requirements follow-up
* To understand the purpose of the trial and willing to sign informed consent and accept clinical follow-up

Exclusion Criteria:

* AMI within 7 days.
* CTO (TIMI 0), the left main lesion, ostial lesion and transplant vascular lesions, the bifurcation lesion (reference collateral blood vessel diameter of 2.5 mm or higher), stent restenosis lesions and to deal with three pathological changes;
* Severe calcified lesion unable to predilate.
* The distortion of the stent was hampered by lesions.
* NYHA≥Ⅲ or LVEF<40%.
* Prior PCI within 1 year.
* Pregnancy or lactation, and planning pregnancy or lactation.
* Subjects have bleeding tendency or blood coagulation dysfunction or PCI contraindications, or anticoagulant therapy taboo or can't continue to take DAPT at least 1 year.
* There are other diseases (such as cancer,malignant tumor ,congestive heart failure,organ transplantation or candidate) or abuse history (alcohol cocaine heroin, etc.), scheme compliance is poor, interference related data explanation or the limited life (< 1 year).
* To aspirin heparin clopidogrel cobalt chromium alloy rapamycin PLA polymer contrast agent of one of allergy.
* Serious liver and kidney function are not complete subject(ALT and AST were three times greater than the upper limit of normal).
* Before enrolling to participate in other clinical trials and not reached the primary endpoint.
* Non-compliant subject and could not finish the trial in accordance with the requirements of the subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will plan for a total of 55 patients with Non ST-ACS (all of the patients was selected in different blood vessels, a total of up to two target disease Variable and each target lesion 1 stents, such as placing stents need more than one in the operation, require the use of EXCEL stents, mix does not recommend the same patients Other brand support, unless save extra stents.) Choose lesions reference diameter of 2.5 mm to 4.0 mm (visual), each lesion length 32 mm or less (visual), participants must conform to the standard can be selected.
Sampling Method: Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Neointimal coverage of EXCEL biodegradable polymer-coated sirolimus-eluting stent | 9 months
  offline OCT analysis will be performed independently by 2 investigators blinded to patient characteristics and to the stent used. Proprietary software will be used to analyze cross-sections at 1-mm intervals(every 5 frames) within the stented segment. In each cross-section, the number of struts was counted. Struts were classified as uncovered if any part of the strut was visibly exposed to the lumen, or covered if a layer of tissue was visible all over the reflecting surfaces.

SECONDARY OUTCOMES:
Major Adverse Cardiovascular of EXCEL biodegradable polymer-coated sirolimus-eluting stent | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: HUILIANG LIU, MD, Study Chair — CHINESE ARMED POLICE FORCE GENRAL HOSPITAL
Locations (1):
- Cardiology Department, Chinese Armed Police Force Genral Hospital, Beijing China, Beijing, China

REFERENCES:
- [Background] Ozaki Y, Okumura M, Ismail TF, Naruse H, Hattori K, Kan S, Ishikawa M, Kawai T, Takagi Y, Ishii J, Prati F, Serruys PW. The fate of incomplete stent apposition with drug-eluting stents: an optical coherence tomography-based natural history study. Eur Heart J. 2010 Jun;31(12):1470-6. doi: 10.1093/eurheartj/ehq066. Epub 2010 Apr 2. PMID 20363765
- [Result] Finn AV, Joner M, Nakazawa G, Kolodgie F, Newell J, John MC, Gold HK, Virmani R. Pathological correlates of late drug-eluting stent thrombosis: strut coverage as a marker of endothelialization. Circulation. 2007 May 8;115(18):2435-41. doi: 10.1161/CIRCULATIONAHA.107.693739. Epub 2007 Apr 16. PMID 17438147
- [Result] Matsumoto D, Shite J, Shinke T, Otake H, Tanino Y, Ogasawara D, Sawada T, Paredes OL, Hirata K, Yokoyama M. Neointimal coverage of sirolimus-eluting stents at 6-month follow-up: evaluated by optical coherence tomography. Eur Heart J. 2007 Apr;28(8):961-7. doi: 10.1093/eurheartj/ehl413. Epub 2006 Nov 29. PMID 17135281
- [Result] Kubo T, Imanishi T, Kitabata H, Kuroi A, Ueno S, Yamano T, Tanimoto T, Matsuo Y, Masho T, Takarada S, Tanaka A, Nakamura N, Mizukoshi M, Tomobuchi Y, Akasaka T. Comparison of vascular response after sirolimus-eluting stent implantation between patients with unstable and stable angina pectoris: a serial optical coherence tomography study. JACC Cardiovasc Imaging. 2008 Jul;1(4):475-84. doi: 10.1016/j.jcmg.2008.03.012. PMID 19356470
- [Result] Stone GW, Maehara A, Lansky AJ, de Bruyne B, Cristea E, Mintz GS, Mehran R, McPherson J, Farhat N, Marso SP, Parise H, Templin B, White R, Zhang Z, Serruys PW; PROSPECT Investigators. A prospective natural-history study of coronary atherosclerosis. N Engl J Med. 2011 Jan 20;364(3):226-35. doi: 10.1056/NEJMoa1002358. PMID 21247313
- [Result] Farb A, Burke AP, Kolodgie FD, Virmani R. Pathological mechanisms of fatal late coronary stent thrombosis in humans. Circulation. 2003 Oct 7;108(14):1701-6. doi: 10.1161/01.CIR.0000091115.05480.B0. Epub 2003 Sep 22. PMID 14504181
- [Result] Guagliumi G, Sirbu V, Musumeci G, Bezerra HG, Aprile A, Kyono H, Fiocca L, Matiashvili A, Lortkipanidze N, Vassileva A, Popma JJ, Allocco DJ, Dawkins KD, Valsecchi O, Costa MA. Strut coverage and vessel wall response to a new-generation paclitaxel-eluting stent with an ultrathin biodegradable abluminal polymer: Optical Coherence Tomography Drug-Eluting Stent Investigation (OCTDESI). Circ Cardiovasc Interv. 2010 Aug;3(4):367-75. doi: 10.1161/CIRCINTERVENTIONS.110.950154. Epub 2010 Jul 20. PMID 20647562